CLINICAL TRIAL: NCT05253651
Title: An Open-label Randomized Phase 3 Study of Tucatinib in Combination With Trastuzumab and mFOLFOX6 Versus mFOLFOX6 Given With or Without Either Cetuximab or Bevacizumab as First-line Treatment for Subjects With HER2+ Metastatic Colorectal Cancer
Brief Title: A Study of Tucatinib With Trastuzumab and mFOLFOX6 Versus Standard of Care Treatment in First-line HER2+ Metastatic Colorectal Cancer
Acronym: MOUNTAINEER-03
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGNTUC-029; C4251008 (Other: Alias Study Number); 2024-514180-25-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Cancer; CRC; Seattle Genetics
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tucatinib; Trastuzumab; Bevacizumab; Cetuximab; Oxaliplatin; Leucovorin; Levoleucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tucatinib Arm (Experimental): Tucatinib + trastuzumab + mFOLFOX6
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: oxaliplatin; Drug: leucovorin; Drug: levoleucovorin; Drug: fluorouracil
- Standard of Care Arm (Active Comparator): Either (1) mFOLFOX6, (2) mFOLFOX6 and bevacizumab, or (3) mFOLFOX6 and cetuximab
  Interventions: Drug: bevacizumab; Drug: cetuximab; Drug: oxaliplatin; Drug: leucovorin; Drug: levoleucovorin; Drug: fluorouracil

INTERVENTIONS:
Drug: tucatinib — 300mg given by mouth (orally) twice daily
  Other Names: TUKYSA, ONT-380, ARRY-380, PF-07265792
  Arms: Tucatinib Arm
Drug: trastuzumab — 8mg/kg loading dose will be given into the vein (IV; intravenously) on Cycle 1 day 1, followed by 6mg/kg given by IV every 3 weeks thereafter.
  Other Names: Herceptin
  Arms: Tucatinib Arm
Drug: bevacizumab — 5mg/kg given by IV every 2 weeks
  Other Names: Avastin
  Arms: Standard of Care Arm
Drug: cetuximab — 400mg/m2 loading dose will be given by IV on Cycle 1 day 1, followed by 250mg/m2 given by IV weekly
  Other Names: Erbitux
  Arms: Standard of Care Arm
Drug: oxaliplatin — 85mg/m2 given by IV every 2 weeks. Component of mFOLFOX6.
Drug: leucovorin — 400mg/ m2 given by IV every 2 weeks. Component of mFOLFOX6.
Drug: levoleucovorin — 200mg/ m2 given by IV every 2 weeks. May be given in place of leucovorin. Component of mFOLFOX6.
Drug: fluorouracil — 400mg/m2 given by IV bolus then 2400mg/m2 given by continuous IV infusion (over 46-48 hours) every 2 weeks. Component of mFOLFOX6.

SUMMARY:
This study is being done to find out if tucatinib with other cancer drugs works better than standard of care to treat participants with HER2 positive colorectal cancer. This study will also determine what side effects happen when participants take this combination of drugs. A side effect is anything a drug does to the body besides treating your disease.

Participants in this study have colorectal cancer that has spread through the body (metastatic) and/or cannot be removed with surgery (unresectable).

Participants will be assigned randomly to the tucatinib group or standard of care group. The tucatinib group will get tucatinib, trastuzumab, and mFOLFOX6. The standard of care group will get either:

* mFOLFOX6 alone,
* mFOLFOX6 with bevacizumab, or
* mFOLFOX6 with cetuximab mFOLFOX6 is a combination of multiple drugs. All of the drugs given in this study are used to treat this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed adenocarcinoma of the colon or rectum which is locally advanced unresectable or metastatic
* Able to provide the most recently available formalin-fixed paraffin-embedded (FFPE) tumor tissue blocks (or freshly sectioned slides) obtained prior to treatment initiation to a central laboratory

  * If archival tissue is not available, a newly-obtained baseline biopsy of an accessible tumor lesion is required within 35 days prior to start of study treatment
* HER2+ disease as determined by a tissue based assay performed at a central laboratory.
* Participant has rat sarcoma viral oncogene homolog wild-type (RAS WT) disease as determined by local or central testing. For central RAS analysis, tissue sample must be analyzed within 1 year of biopsy date.
* Radiographically measurable disease per RECIST v1.1 with:

  * At least one site of disease that is measurable and that has not been previously irradiated, or
  * If the participant has had previous radiation to the target lesion(s), there must be evidence of progression since the radiation
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* CNS Inclusion - based on contrast brain magnetic resonance imaging, participants may have any of the following:

  * No evidence of brain metastases
  * Previously treated brain metastases which are asymptomatic

Exclusion Criteria:

* Prior systemic anticancer therapy for colorectal cancer (CRC) in the locally advanced unresectable or metastatic setting; note that participants may have received a maximum of 2 doses of mFOLFOX6 in the locally advanced/unresectable or metastatic setting prior to randomization.

  * Note: May have received chemotherapy for CRC in the adjuvant setting if it was completed >6 months prior to enrollment
* Radiation therapy within 14 days prior to enrollment (or within 7 days in the setting of stereotactic radiosurgery)
* Previous treatment with anti-HER2 therapy
* Ongoing Grade 3 or higher neuropathy
* Active or untreated gastrointestinal (GI) perforation at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2026-04-03 (Estimated); Study Completion 2029-07-27 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) by Blinded Independent Central Review (BICR) | Up to approximately 3 years
  The time from the date of randomization to the BICR assessment of disease progression according to RECIST v1.1 or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 6 years
  The time from randomization to death from any cause
Confirmed objective response rate (cORR) per RECIST v1.1 by BICR | Up to approximately 3 years
  The proportion of participants with confirmed complete response (CR) or partial response (PR) according to RECIST v1.1, as assessed by BICR
PFS per RECIST v1.1 by investigator assessment | Up to approximately 3 years
  The time from the date of randomization to the investigator assessment of disease progression according to RECIST v1.1 or death from any cause
cORR per RECIST v1.1 by investigator assessment | Up to approximately 3 years
  The proportion of participants with confirmed CR or PR according to RECIST v1.1, as assessed by investigators
Duration of response (DOR) per RECIST v1.1 by BICR | Up to approximately 3 years
  The time from first documentation of objective response (CR or PR that is subsequently confirmed) to the first documentation of disease progression per RECIST v1.1 or death from any cause
DOR per RECIST v1.1 by investigator assessment | Up to approximately 3 years
  The time from first documentation of objective response (CR or PR that is subsequently confirmed) to the first documentation of disease progression per RECIST v1.1 or death from any cause
Time to second progression or death (PFS2) | Up to approximately 3 years
  The time from randomization to disease progression on the next-line of therapy, or death from any cause
Incidence of adverse events (AEs) | Through 30 days after the last study treatment; approximately 1 year
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Incidence of dose alterations | Through 30 days after the last study treatment; approximately 1 year
Trough concentration (Ctrough) | Approximately 4 months
  PK parameter
Change from baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQC30) score | Through 30-37 days after the last study treatment; approximately 1 year
  Change from baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) scores. Scale scores range from 0-100. For functioning and global health status/quality of life (QoL) scales, higher scores indicate better functioning or global health status/quality of life (QoL). For symptom scales, higher scores indicate greater symptom burden.
Time to meaningful change in EORTC QLQ30 score | Through 30-37 days after the last study treatment; approximately 1 year
  The time from baseline to the first onset of a ≥10-point changes in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) scores. Scale scores range from 0-100.
  For functioning and global health status/QoL scales, higher scores indicate better functioning or global health status/QoL. For symptom scales, higher scores indicate greater symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (373):
- United States (126):
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - Mayo Clinic Building - Phoenix, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Los Angeles Cancer Network - Anaheim, Anaheim, California
  - Kaiser Permanente Anaheim Kraemer Medical Offices, Anaheim, California
  - Kaiser Permanente Baldwin Park Medical Center, Baldwin Park, California
  - Kaiser Permanente Bellflower Medical Offices, Bellflower, California
  - Kaiser Permanente Fontana Medical Center, Fontana, California
  - Los Angeles Cancer Network - Fountain Vally, Fountain Valley, California
  - Los Angeles Hematology Oncology Medical Group, Glendale, California
  - Kaiser Permanente South Bay Medical center, Harbor City, California
  - Kaiser Permanente Alton/Sand Canyon Medical Offices, Irvine, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - USC Norris Koreatown - Medical Oncology, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Offices, Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles Medical Center, Los Angeles, California
  - USC Norris Oncology/Hematology - Newport Beach, Newport Beach, California
  - Kaiser Permanente Ontario Medical Center, Ontario, California
  - Kaiser Permanente Panorama City Medical Center, Panorama City, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Los Angeles Hematology Oncology Medical Group, Pasadena, California
  - Kaiser Permanente Riverside Medical Center, Riverside, California
  - Kaiser Permanente San Diego Mission Road (Regulatory and Lab Supplies), San Diego, California
  - Kaiser Permanente Zion Medical Center, San Diego, California
  - Kaiser Permanente San Marcos Medical Offices, San Marcos, California
  - Los Angeles Hematology Oncology Medical Group, Van Nuys, California
  - Kaiser Permanente Woodland Hills Medical Center, Woodland Hills, California
  - Rocky Mountain Cancer Centers, LLP, Aurora, Colorado
  - Rocky Mountain Cancer Centers, LLP, Boulder, Colorado
  - Rocky Mountain Cancer Centers, LLP, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - Rocky Mountain Cancer Centers, LLP, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, LLP, Littleton, Colorado
  - Rocky Mountain Cancer Centers, LLP, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, LLP, Longmont, Colorado
  - Rocky Mountain Cancer Centers, LLP, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, LLP, Thornton, Colorado
  - Mount Sinai Medical Center Aventura ER, Aventura, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Alliance for Multispecialty Research LLC., Merriam, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Cancer Institute - Downtown, Louisville, Kentucky
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Norton Audubon Hospital, Louisville, Kentucky
  - Norton Cancer Institute, Audubon Hospital Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital, Louisville, Kentucky
  - Norton Cancer Institute, Brownsboro Hospital Campus, Louisville, Kentucky
  - Minnesota Oncology Hematology, PA, Burnsville, Minnesota
  - Allina Health Cancer institute, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology, PA, Coon Rapids, Minnesota
  - M Health Fairview Cancer Clinic-Edina, Edina, Minnesota
  - Minnesota Oncology Hematology, PA, Edina, Minnesota
  - Minnesota Oncology Hematology, PA, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA, Maple Grove, Minnesota
  - M Health Fairview St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA, Maplewood, Minnesota
  - Allina Health Cancer Institute (Virginia Piper Cancer Institute), Minneapolis, Minnesota
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Health Cancer Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center Outpatient Pharmacy, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Regulatory Location: MMCORC, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Allina Health Cancer Institute-United(VPCI), Saint Paul, Minnesota
  - Minnesota Oncology Hematology, PA Cornerstone Medical Specialty Center, Woodbury, Minnesota
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - MSK Bergen, Montvale, New Jersey
  - MSK Commack, Commack, New York
  - MSK Westchester, Harrison, New York
  - Rockefeller Outpatient Pavilion (53rd Street), New York, New York
  - Memorial Solan Kettering Cancer Center- Main Campus, New York, New York
  - MSK Nassau, Uniondale, New York
  - Duke University Hospital, Durham, North Carolina
  - Duke University Medical Center, Duke Cancer Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - FirstHealth Cancer Center, Pinehurst, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Oncology and Hematology Care Clinic - Westside, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - UPMC Hillman Cancer Center - Beaver, Beaver, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Hillman Cancer Center at Arnold Palmer Pavilion, In Partnership with Excela Health, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center - Pinnacle (Community Osteopathic / Medical Sciences Pavillion), Harrisburg, Pennsylvania
  - UPMC Hillman Cancer Center at Arnold Palmer Pavilion, In Partnership with Excela Health, Irwin, Pennsylvania
  - UPMC Hillman Cancer Center - Pinnacle (Ortenzio Cancer Center), Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - St Margarets, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC)/Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant (HOA), Pittsburgh, Pennsylvania
  - St. Clair Cancer Center Medical Oncology, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center - Washington, Washington, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center(IPC), Irving, Texas
  - Oncology & Hematology Associates of Southwest Virginia, Inc. D.B.A Blue Ridge Cancer Care, Blacksburg, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Low Moor, Virginia
  - Oncology & Hematology Associates of Southwest Virginia Inc dba Blue Ridge Cancer Care, Roanoke, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc. D.B.A Blue Ridge Cancer Care, Salem, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Wytheville, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Providence Regional Medical Center Everett, Everett, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
- Argentina (6):
  - Centro de Investigacion Pergamino SA, Pergamino, Buenos Aires
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - Instituto Medico Especializado Alexander Fleming, Buenos Aires
  - Hospital Britanico de Buenos Aires, CABA
  - IONC Instituto Oncologico de Cordoba Fundacion Richardet Longo, Córdoba
  - CEMAIC - Centro Medico Privado, Córdoba
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - St Vincent's Hospital, Fitzroy, Victoria
- Austria (5):
  - Klinikum Wels-Grieskirchen GmbH Austria, Wels, Upper Austria
  - Landesapotheke Salzburg, Salzburg
  - Uniklinikum Salzburg, Landeskrankenhaus, Salzburg
  - Klinikum Wels-Grieskirchen GmbH Austria, Wels
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Belgium (8):
  - Institut Jules Bordet, Anderlecht
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZA, Edegem
  - CHU HELORA - Hopital de Jolimont, Haine-Saint-Paul
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Chretien - Clinique MontLegia, Liège
  - Maag-,Darm- en Leverziekten AZ Turnhout, Turnhout
  - Oncologisch Dagziekenhuis AZ Turnhout Campus Sint-Elisabeth, Turnhout
- Brazil (9):
  - CIONC-Centro Integrado de Oncologia de Curitiba, Curitiba, Paraná
  - Instituto De Educação, Pesquisa e Gestão em Saúde - Instituto Américas, Barra da Tijuca, Rio de Janeiro
  - Institute de Educacao, Pesquisa e Gestao em Saude - Instituto COI, Rio de Janeiro, Rio de Janeiro
  - Centro Integrado de Pesquisa em Oncologia CIPO-GHC / Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos/Fundacao Pio XII, Barretos, São Paulo
  - Centro de Pesquisas Clinicas da Fundação Doutor Amaral Carvalho, Jaú, São Paulo
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia., Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira., São Paulo
- Canada (5):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Chile (3):
  - Oncocentro Apys, Viña del Mar, Región de Valparaíso
  - Biocenter, Concepción
  - Centro de estudios clinicos SAGA, Santiago
- China (30):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The 900th Hospital of The Chinese People's Liberation Army Joint Logistics Support Force, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The Sixth Affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Meizhou People's hospital, Meizhou, Guangdong
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Nanyang Second General Hospital, Nanyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - LinYi Cancer Hospital, Linyi, Shandong
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Province Cancer Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - Army Specialty Medical Center of The Chinese People's Liberation Army, Chongqing
  - Shanghai General Hospital, Shanghai
- France (21):
  - Centre Hospitalier Regional et Universitaire de Besancon - Hopital Jean-Minjoz, Besançon, Other
  - Institut Sainte Catherine, Avignon
  - CHU Brest Hopital Cavale Blanche, Brest
  - CHU Estaing, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - Center Georges-Francois Leclerc, Dijon
  - Hopital Edouard Herriot, Lyon
  - Höpital Saint-Joseph, Marseille
  - Centre Hospitalier Universitaire Nantes-Hotel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital Saint-Louis, Paris
  - Pharmacy Address:Hopital Saint-Louis, Paris
  - Hopital Saint-Antoine, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - CHU Bordeaux Hopital Haut Leveque, Pessac
  - CHU Poitiers, Poitiers
  - CHU de Rouen, Rouen
  - Institut de Cancérologie de l'Ouest - Saint-Herblain, Saint-Herblain
  - Centre Hospitalier Universitaire Sainte-Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Institut de Cancerologie Strasbourg Europe, Strasbourg
  - CHU Toulouse-Rangueil, Toulouse
- Germany (21):
  - CCC Muenchen TUM, Munich, Bavaria
  - LMU Klinikum - Campus Großhadern, München, Bavaria
  - Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Landesdirektion Sachsen Dienststelle Leipzig, Leipzig, Saxony
  - Klinikum St. Marien Amberg, Amberg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Apotheke Johannstadt, Dresden
  - Gemeinschaftspraxis Hämatologie - Onkologie, Dresden
  - Technische Universität Dresden, Medizinische Fakultät Carl Gustav Carus, Dresden
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Hämatologisch Onkologische Praxis Eppendorf (HOPE), Hamburg
  - ZytoService Deutschland GmbH, Hamburg
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - Asklepios Tumorzentrum Hamburg, Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Rechts der Isar der Technischen Universitaet Muenchen, München
  - Klinikum rechts der Isar der TU München, Krankenhausapotheke, München
  - Universitaetsklinikum Ulm, Ulm
- Greece (5):
  - Athens Medical Center - Psychikon branch, Athens, Attikí
  - University General Hospital "Attikon", Athens, Chaidari
  - "University General Hospital of Heraklion Oncology Unit ", Heraklion, Crete
  - "Papageorgiou" General Hospital of Thessaloniki 2nd Internal Medicine/Oncology Clinic of Aristotle, Nea Efkarpia, Thessaloniki
  - Evgenidion Clinic Agia Trias Oncology Department, Athens
- Ireland (7):
  - Cork University Hospital,Department of Medical Onncology, Cork
  - Bon Secours Hospital, Cork
  - St Vincents University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - Beaumont Hospital, Dublin
  - University Hospital Waterford, Waterford
- Italy (31):
  - Azienda Ospedaliera Universitaria Cagliari, Monserrato, Cagliari
  - Farmacia AOU Cagliari - Presidio Ospedaliero ' Duilio Casula' di Monserrate, Monserrato, Cagliari
  - UOC Oncologia Medica - Dipartimento Onco Ematologico AORN San Giuseppe Moscati di Avellino, Avellino, Campania
  - IRCCS Ospedale Policlinico San Martino Farmacia, Genova, GE
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - UOC Oncologia, Azienda Ospedaliera Cardinale Giovanni Panico, Tricase, Lecce
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - lstituto Europeo di Oncologia, Milan, Lombardy
  - Niguarda Cancer Center Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - UMaCA U.O.S.D. Farmacia Ospedaliera, Napoli, Naples
  - IRCCS Ospedale Policlinico San Martino, Genova, Other
  - Ospedale S Chiara Farmacia, Pisa, Other
  - Servizio Farmacia Azienda Ospedaliera Universitaria lntegrata (AOUI) di Verona, Verona, Other
  - Farmacia Sperimentazioni, Reggio Emilia, RE
  - UOC Oncologia Medica, ARNAS GARIBALDI - PRESIDIO OSPEDALIERO NESIMA, Catania, Sicily
  - SODc Oncologia Medica e Clinica, AOU Careggi, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
  - Struttura Semplice Dipartimentale di Oncologia Medica e Terapia Biomolecolare Azienda Ospedaliero, Foggia
  - lstituto Europeo di Oncologia Servizio Farmacia, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori Farmacia, Milan
  - Istituto Oncologico Veneto-IRCCS Farmacia, Padua
  - Fondazione IRCCS Policlinico San Matteo Farmacia, Pavia
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Farmacia UFA, Reggio Emilia
  - S.C Oncologia Arcispedale Santa Maria Nuova, Reggio Emilia
  - Farmacia degli Sperimentali Policlinico Gemelli IRCCS, Roma
  - ASST della Valtellina e dell'alto Lario - Presidio Ospedaliero di Sondrio, Sondrio
  - ASST della Valtellina e dell'alto Lario- Presidio Ospedaliero di Sondrio Farmacia, Sondrio
  - U.O.C. Oncologia Azienda Ospedaliera Universitaria lntegrata (AOUI) di Verona, Verona
- Japan (17):
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - St. Marianna University Hospital, Kawasaki-shi, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Osaka General Medical Center, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-shi, Osaka
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - National Hospital Organization Osaka National Hospital, Osaka
- Netherlands (5):
  - St. Antonius Hospital, Nieuwegein, Other
  - Netherlands Cancer Institute, Amsterdam
  - Klinische Farmacie, Nieuwegein
  - St. Antonius Ziekenhuis - Ziekenhuis Utrecht, Utrecht
  - Viecuri Medisch Centrum, Venlo
- Norway (3):
  - Sjukehusapoteket i Bergen [Bergen Hospital Pharmacy], Bergen
  - Helse Bergen HF, Haukeland University Hospital, Bergen
  - Oslo University Hospital (OUH) - The Norwegian Radium Hospital, Oslo
- Poland (9):
  - Przychodnia Lekarska KOMED Roman Karaszewski, Konin, Greater Poland Voivodeship
  - Narodowy lnstytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy lnstytut Badawczy, Warsaw, Masovian Voivodeship
  - Marii Sklodowskiej-Curie Panstwowy lnstytut Badawczy, Warsaw, Masovian Voivodeship
  - Wojskowy Instytut Medyczny Klinika Onkologii, Warsaw, Masovian Voivodeship
  - Wojskowy Instytut Medyczny, Warsaw, Masovian Voivodeship
  - MRUK-MED | Sp. z.o.o Apteka szpitalna, Rzeszów, Podkarpackie Voivodeship
  - MRUK-MED | Sp. z.o.o, Rzeszów, Podkarpackie Voivodeship
  - Apteka Szpitalna Uniwersytie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Salve Medica Apteka Szpitalna, Lodz
- Portugal (4):
  - Hospital Garcia de Orta, Almada
  - Unidade Local de Saude da Guarda-Hospital Sousa Martins, Guarda
  - Fundacao Champalimaud, Lisbon
  - Centro Hospitalar Universitário de Santo Antonio,E.P.E., Porto
- Narodny Onkologicky ustav II.Onkologicka Klinika LFUK a NOU, Bratislava, Slovakia
- South Korea (7):
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (26):
  - Hospital Duran i Reynals - Institut Catala d'Oncologia L'Hospitalet (ICO L'Hospitalet), L'Hospitalet de Llobregat, Barcelona
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - CETIR Viladomat, Barcelona, Other
  - Complejo Hospitalario Universitario de Canarias, San Cristóbal de La Laguna, Santa CRUZ DE Tenerife
  - Hospital General Universitario de Alicante, Alicante
  - Radiology: CETIR Ascires, Barcelona
  - Data review: Vall d'Hebron institute of Oncology (VHIO)., Barcelona
  - Hospital Vall d'Hebron Unidad de Farmacia de Ensayos Clinicos Oncohematologia, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Clínica Universidad de Navarra (Madrid), Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga (Hospital Civil), Málaga
  - Complejo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Quiron Salud Zaragoza, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (4):
  - Pharmacy:Kantonsspital Winterthur, Winterthur, Other
  - Zuripharm AG, Schlieren
  - Kantonsspital Winterthur, Winterthur
  - Universitatsspital Zurich - Klinik fur Medizinische Onkologie und Hamatologie USZ, Zurich
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Hospital Clinical Trial Pharmacy, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital LinKou, Taoyuan District
- United Kingdom (11):
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Chelsea
  - The Royal Marsden Hospital, Sutton, Surrey
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Oncology Centre, Cambridge
  - Leeds Teaching Hospitals NHS Trust, st James's Institute of Oncology, Leeds
  - Guy's and Saint Thomas' NHS Foundation Trust, London
  - The Royal Marsden Hospital - Chelsea Site, London
  - The Royal Marsden NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Strickler JH, Bekaii-Saab T, Cercek A, Heinemann V, Nakamura Y, Raghav K, Siena S, Tabernero J, Van Cutsem E, Yoshino T, Ramos J, Guan X, Andre T. MOUNTAINEER-03 phase III study design: first-line mFOLFOX6 + tucatinib + trastuzumab for HER2+ metastatic colorectal cancer. Future Oncol. 2025 Feb;21(3):303-311. doi: 10.1080/14796694.2024.2441101. Epub 2024 Dec 26. PMID 39723627
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNTUC-029